CLINICAL TRIAL: NCT04259645
Title: Volume Versus Concentration: A Prospective, Double Blind, Parallel Study to Compare the Clinical Effectiveness of Single Shot Quadratus Lumborum Block Using Either a High Volume/Low Concentration or Low Volume/High Concentration Injectate for Total Hip Arthroplasty.
Brief Title: Volume Versus Concentration: Clinical Effectiveness of Single Shot Quadrates Lumborum Block Using Either a High Volume/Low Concentration or Low Volume/High Concentration Injectate for Total Hip Arthroplasty.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anna Uskova (Other)
Responsible Party: Sponsor-Investigator, Anna Uskova, Clinical Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY19090192
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Acute Pain
Keywords: Hip; Anesthesia,conduction; arthroplasty
MeSH Terms: conditions — Acute Pain | interventions — Bupivacaine; Hospitals, Low-Volume; Hospitals, High-Volume

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a prospective, randomized, double blinded, parallel trial at the University of Pittsburgh Medical Center (UPMC) Shadyside Hospital.
Who Masked: Participant, Outcomes Assessor
Masking Description: An envelope will contain the randomized concentration and volume of ropivacaine to be administered to the patient. Once the anesthesiologist knows which volume he is going to administer, he will reseal the envelope and return it to the research team. This process will allow only the anesthesiologist performing the block to have knowledge of the volume he is administering, keeping both the patients and outcome assessor of the research team blinded.
  The anesthesiologist will fill the syringe with the appropriate volume of medication. Immediately after, he will cover the numbers on the syringe with a piece of opaque tape, preventing any others from visualizing the volume to be administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Volume group (Active Comparator): 30 subjects randomized to Low Volume will receive unilateral Quadratus Lumborum block type II. Each subject received 20mL Bupivacaine 0.375%.
  Interventions: Drug: Drug: Bupivacaine 0.375% diluted to 0.1875%
- High Volume group (Experimental): 30 subjects randomized to High Volume will receive unilateral Quadratus lumborum block Type II. Each subject was given 20mL Bupivacaine 0.375% diluted with 20mL normal saline to total 40mL (concentration decreased by half - 0.1875%).
  Interventions: Drug: Drug: Bupivacaine 0.375% 20 mL

INTERVENTIONS:
Drug: Drug: Bupivacaine 0.375% 20 mL — 20 mL 0.375% Bupivacaine
  Other Names: Low Volume
  Arms: High Volume group
Drug: Drug: Bupivacaine 0.375% diluted to 0.1875% — Each block of 0.375% Bupivacaine x 20 ml mixed (diluted) with Normal Saline Solution 20 mL (total 40 mL)
  Other Names: High Volume
  Arms: Low Volume group

SUMMARY:
There is Controversy about what is more critical volume or concentration to achieve an optimum analgesic treatment with quadratus lumborum block. From the experiences of the authors, the regular dose of 20 ml of Bupivacaine at 0.375% concentration could not be enough in some cases to produce an optimum analgesic treatment, especially in hip arthroplasties. What is proposed in this study is to evaluate whether the volume injected in the quadratus lumborum block is more important than the concentration of the local anesthetic in terms of control of pain during the next 24 hours after surgery and opioid consumption.

DETAILED DESCRIPTION:
The Quadratus Lumborum Block (QLB) was originally described by Blanco in 2007 as a posterior variation of the Transversus Abdominis Plane block. It is now, however, recognized as a unique, alternative, and separate interfascial plane block. The QLB has been studied and compared with other types of blocks and it may offer several advantages such as simplicity, safety, and avoidance of hypotension. Additionally, dermatomal coverage may be greater than for other types of blocks. In cadaveric studies the paravertebral spread of dye was found from T7-L5 , although an vivo study in healthy volunteers showed the paravertebral spread of the contrast solution only between T10-L1 at 1 hour after the block. It is noted that while these anatomical studies invariably show the spread of contrast or dye extending to the paravertebral space that spread may be limited in degree. Thus follows a point of significant controversy as to whether the paravertebral space is in fact the block's primary site of action or whether it acts primarily on nerves, radicular and sympathetic, situated in the thoracolumbar fascia. Questions of mechanism and site of action notwithstanding, the safety and clinical efficacy of this block has been clearly demonstrated in multiple types of surgeries including abdominal laparoscopic , open laparotomy , urologic , and general surgery with analgesia lasting roughly 24 hours, decreased consumption of opioids, decreased time to ambulation, and decreased hospital length of stay. In recent studies, QL block employment was shown to produce a significant reduction in length of stay during hip surgery as well as similar analgesia to Lumbar Plexus blockade.

The quadratus lumborum block has since 2016 become standard of care for abdominal and hip surgeries at our institution, replacing paravertebral and lumbar plexus blocks respectively, and as part of a broader multimodal analgesia institutional ERAS (Enhanced Recovery After Surgery) protocol. Coincident with its implementation we have seen significant reductions in opiate and PCA use as well as hospital length of stay. Similar results have been reported by other institutions.

Since the first description of this technique, several approaches to and anatomic targets within the quadratus lumborum plane have been described although their mechanism of action, spread, and relative clinical effectiveness remain areas of some debate. There remain many unanswered questions regarding this block and its subtypes. It is, for example, unknown if one technique would be better than another for different types of surgery. Likewise little is known of the relative importance of local anesthetic concentration and injectate volume - the principal question addressed by this proposed study.

ELIGIBILITY:
Inclusion Criteria:

Patients 18-80 years old Patients undergoing total hip arthroplasty BMI 19-45, >50 kg Male and Female All races American Society of Anesthesiologists physical status classification I, II, III Spinal Anesthesia Provided

Exclusion Criteria:

Pregnancy Non english speaking or inability to participate in the study Patients with coagulopathy or With INR >1.5 the day of the surgery. pharmacologic coagulopathy: patients on xarelto, plavix, or any kind of "Blood Thinners" Chronic steroid use: patients with consumption of steroid for more than 3 months.

Chronic pain: pain for more than 3 months Chronic opiate use : consumption of opioids for more than 3 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Uskova, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of pittsburgh, Pittsburgh, Pennsylvania
  - UPMC shadyside hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Volume Group: 30 subjects randomized to Low Volume will receive unilateral Quadratus Lumborum block type II. Each block of 0.375% Bupivacaine x 20 ml
  Drug: Bupivacaine 0.375%: Each block of 0.375% Bupivacaine x 20 ml
- High Volume Group: 30 subjects randomized to High Volume will receive unilateral Quadratus lumborum block Type II. Each block of 0.375% Bupivacaine x 20 mL + Normal Saline Solution 20 mL
  Drug: Bupivacaine 0.375% Bupivacaine x 20 mL + Normal Saline Solution 20 mL (total 40mL)
Period: Overall Study
Arm/Group | Low Volume Group | High Volume Group
Started | 29 | 31
Completed | 29 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- High Volume Group: 30 subjects randomized to High Volume will receive unilateral Quadratus lumborum block Type II. Each block of 0.375% Bupivacaine x 20 mL + Normal Saline Solution 20 mL
  Drug: Bupivacaine 0.375% 20 mL: Each block of 0.375% Bupivacaine x 20 mL diluted with 20mL of Normal Saline Solution
- Total: Total of all reporting groups
Arm/Group | Low Volume Group | High Volume Group | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.1) | 65.4 (8.7) | 64.55 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 16 | 16 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 60
BMI [Mean (Standard Deviation); unit: kg/m2] | 31.0 (5.4) | 30.6 (5.7) | 30.8 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Consumption of Opioids During the First 24 Hours After Surgery.
Description: Opioids administered to the patient in 24 hours, measured as averaged morphine milligram equivalent
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg morphine equivalents per 24 hours
Groups:
- Low Volume Group: 30 subjects randomized to Low Volume will receive unilateral Quadratus Lumborum block type II. Each block of 0.375% Bupivacaine x 20 ml
- High Volume Group: 30 subjects randomized to High Volume will receive unilateral Quadratus lumborum block Type II. Each block of 0.375% Bupivacaine x 20 mL + Normal Saline Solution 20 mL
Arm/Group | Low Volume Group | High Volume Group
Number analyzed (Participants) | 29 | 31
mg morphine equivalents per 24 hours | 46.2 (25.9) | 35.0 (27.1)

2. Primary Outcome: Pain Measurement Through VAS (Visual Analogue Score) at Rest
Description: pain scores at rest at 3 hours after surgery (minimum 0 - maximum 10)
Time Frame: 3-hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Volume Group | High Volume Group
Number analyzed (Participants) | 29 | 31
score on a scale | 4.52 (2.76) | 4.48 (2.81)

3. Primary Outcome: Pain Measurement Through VAS (Visual Analogue Score) at Rest
Description: pain scores at rest at 6 hours after surgery (minimum 0 - maximum 10)
Time Frame: 6-hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Volume Group | High Volume Group
Number analyzed (Participants) | 29 | 31
score on a scale | 5.76 (2.71) | 5.08 (2.21)

4. Primary Outcome: Pain Measurement Through VAS (Visual Analogue Score) at Rest
Description: pain scores at rest at 12 hours after surgery (minimum 0 - maximum 10)
Time Frame: 12-hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Volume Group | High Volume Group
Number analyzed (Participants) | 29 | 31
score on a scale | 5.52 (2.23) | 5.59 (2.83)

5. Primary Outcome: Pain Measurement Through VAS (Visual Analogue Score) at Rest
Description: pain scores at rest at 24 hours after surgery (minimum 0 - maximum 10)
Time Frame: 24-hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Volume Group | High Volume Group
Number analyzed (Participants) | 29 | 31
score on a scale | 4.78 (2.53) | 5.50 (2.75)

6. Secondary Outcome: Time to 100ft Ambulation After Surgery
Description: Time to ambulation after surgery (ability to walk 100 feet).
Time Frame: Post-operative 12-32 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Low Volume Group | High Volume Group
Number analyzed (Participants) | 29 | 31
minutes | 1534 (1055) | 1178 (1219)

7. Secondary Outcome: Time to Consumption of the First Opioid After Surgery.
Description: Time to consumption of the first opioid after surgery.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Low Volume Group | High Volume Group
Number analyzed (Participants) | 29 | 31
minutes | 120 (97) | 165 (270)

8. Secondary Outcome: Time to Hospital Discharge
Description: Time to hospital discharge following surgery, measured in minutes
Time Frame: Post-operative day 1 to post-operative day 5
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Low Volume Group | High Volume Group
Number analyzed (Participants) | 29 | 31
minutes | 1865 (1480) | 1560 (1491)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up until the time of patient discharge, roughly 24-hours.
Arm/Group | Low Volume Group | High Volume Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 0/29 | 0/31

LIMITATIONS AND CAVEATS:
This was a single hospital trial, and external validity may be attenuated. THA is a relatively standardized procedure with similar patient care in the operating room, PACU, and floor ward. With only 60 patients total, this study is underpowered, and the wide standard deviations suggest a need for a much larger study.

Pain score reported as the worst score over the previous 3 hours (interval) and reflects pain at rest post PT activity as day progresses, what may decrease the accuracy of report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT04259645/Prot_SAP_003.pdf
  • Informed Consent Form (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT04259645/ICF_004.pdf